CLINICAL TRIAL: NCT04246632
Title: Prospective, Open Label, Pilot Study of the CapsoCam® Colon Capsule Endoscope (CCE) Compared to Colonoscopy (OC)
Brief Title: CapsoCam® Colon Capsule Endoscope (CCE) Compared to Colonoscopy (OC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capso Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLN-CVI-5248
Record Dates: First submitted 2020-01-24; First posted 2020-01-29 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Intervention Model Description: Multi-Center; Prospective, Open Label, Non-Significant Risk, Pilot Study
Masking Description: PI is masked to Capsule results and capsule reader is masked to colonoscopy results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Open label (Experimental): Single arm study, all subjects receive device
  Interventions: Device: CapsoCam Colon Capsule Endoscopy

INTERVENTIONS:
Device: CapsoCam Colon Capsule Endoscopy — CapsoCam® Colon is intended to provide visualization of the colon and the detection of colon polyps in adults.

SUMMARY:
This non-significant risk pilot study is designed to evaluate safety and performance of the CapsoCam® Colon capsule endoscope in patients who meet the eligibility criteria and are scheduled for colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 50 and 75 years old
2. Subject meets at least one of the following criteria for increased risk for polyps:

   1. Recent history (within 6 months) of positive FIT/iFOBT or Cologuard test
   2. Older than 55 years of age, without prior history of colonoscopy
   3. Has had a positive colonoscopy ≥ 5 years prior to screening visit
   4. And/or having at least two of the following risk factors:

      * Current smoker
      * BMI of ≥30
      * Family history (blood relative) of colorectal cancer
      * Sedentary lifestyle
      * Low fiber/ high fat diet
3. No contraindication for capsule endoscopy or colonoscopy
4. Committed to undergo a colonoscopy, independent of this study within 8 weeks of Capsule ingestion
5. Choose to participate and must have signed the IRB-approved informed-consent document and agreed to release colonoscopy images and results report to Sponsor

Exclusion Criteria:

1. History of negative colonoscopy within the last 10 years
2. History of incomplete colonoscopy
3. Impaired cardiac function assessed as greater than NYHA Class II
4. History of small- or large-bowel obstructive condition
5. Known history of Crohn's disease, swallowing disorder, ulcerative colitis, ischemic bowel disease and/or radiation enteritis
6. Known history of NSAID enteropathy and stricture resulting from taking NSAIDs on a regular basis that, in the opinion of the Investigator, would put the patient at greater risk for capsule endoscope retention
7. Unable to follow or tolerate fasting, bowel preparation, and other study procedures
8. Known allergy to ingredients used in bowel preparation and boosters
9. Daily and/or regular use of narcotics
10. Known or suspected AIDS
11. Uncompensated cirrhosis
12. Prior abdominal radiation therapy
13. Diagnosis of anorexia or bulimia
14. History of or suspicion for: strictures, volvulus or intestinal obstruction; internal hernias or abdominal surgeries that the Investigator considers as an exclusion
15. Known or suspected megacolon
16. Scheduled to undergo MRI examination within 7 days after ingestion of the capsule
17. Has known slow gastric-emptying time or confirmed diagnosis of gastroparesis
18. Pregnant or nursing or is of child-bearing potential and does not practice medically acceptable methods of contraception. Women of childbearing potential (WOCBP) must have a negative urine pregnancy test at screening.
19. Any documented medical or psychological condition or significant concurrent illness which, in the Investigator's opinion, would make it unsafe for the subject to participate in this research study
20. Are currently enrolled in, or participated in within the last 30 days, another clinical study
21. Chronic constipation as defined by <3 bowel movements per week for at least 3 months prior to Screening, or the use of routine laxatives (other than fiber) to attain r regular bowel movements for at least 3 months prior to Screening
22. History of diabetes in which the prolonged fasting schedule could impose additional safety risks, as determined by the investigator

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-01-25 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Efficacy Assessments | Day 1
  Determine the Accuracy of CapsoCam® to detect and measure size of colon polyps relative to the colonoscopy procedure.

SECONDARY OUTCOMES:
Safety Assessments: Incidence of device related serious adverse events (SAEs) and unanticipated adverse device effects (UADEs) | Day 1-3
  All adverse events including SAEs/UADEs will be assessed at all visits. Incidence of serious adverse events (SAEs) and unanticipated adverse device effects (UADEs) will be reported. A serious adverse event is one that meets the definition outlined in Section 8 of this protocol.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Silicon Valley Research Institute, Inc., San Jose, California
  - CapsoVision Research Clinic, Saratoga, California
  - West Michigan Clinical Research Center, Wyoming, Michigan

IPD SHARING:
Plan to Share IPD: No
All IPD will be kept confidential. Safety events/concerns will be shared will all sites without exposing PHI.